CLINICAL TRIAL: NCT05520229
Title: The Evaluation of a Preoperative Anaesthesia Assessment Clinic on Elective Patients After Partial Excision of the Intestine
Brief Title: The Evaluation of a Preanaesthesia Assessment Clinic
Status: Not yet recruiting | Type: Observational
Sponsor: University of Agder (Other)
Collaborators: Sorlandet Hospital HF (Other Government)
Responsible Party: Principal Investigator, Eirunn Wallevik Kristoffersen, Principal Investigator, University of Agder
Other Study IDs: Eirunn W. Kristoffersen
Record Dates: First submitted 2022-08-25; First posted 2022-08-29 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Preoperative Anaesthesia Clinic; Cancellation Rate; Intraoperative Events; Colon Disease
Keywords: Anesthesia, cancellation, pre-operative, clinic, assessment
MeSH Terms: conditions — Colonic Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Pre- Preanaesthesia assessment clinic: Patients who have been to surgery for an elective laparoscopic or open partial intestine from 2014-2017.
- Post- Preanaesthesia assessment clinic: Patients who have been to surgery for an elective laparoscopic or open partial intestine from 2017 and have attended a preanesthesia clinic.

SUMMARY:
International evidence highlights the preanaesthetic assessment clinics (PAC) as a system of benefits for both the patient and the anaesthesiologist. The system has gained global acceptance as a routine method of optimising patients' medical conditions prior to surgery and therefore minimising surgery cancellations and improving hospital efficiency. However, a systematic review found no evidence of the efficiency of (PAC) and therefore we wanted to investigate this with the use of hospitals journals.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the incidence, causes, and consequences of cancellations, and unanticipated intraoperative events after open or laparoscopic surgery of hemicolectomy patients before and after the implementation of a preoperative anaesthesia assessment clinic (PAC).

The primary outcome is to evaluate the incidence of cancellations and unanticipated intraoperative events after open or laparoscopic surgery of hemicolectomy patients before and after implementation of the preoperative anaesthesia assessment clinic (PAC).

The secondary outcome is to evaluate the patients' characteristics, the main events leading to cancellations and the consequences this brings to the patient and the hospital.

Adverse events reported pre-and post-intervention will be analysed. Patient characteristics will be collected: age, gender, diagnosis, reason and type of surgery, patient admission, assessed in PAC or not, ASA classification (American Society of Anesthesiologist Classification system), who performed the assessment (anaesthetic nurse or anaesthesiologist), type of anaesthesia, former diagnosis/disease with impact on anaesthesia/surgery, present smoker, allergies, blood samples, other examinations, cancellation of surgery, reasons and consequences for cancellations, time of anaesthetic assessment before surgery, intraoperative events, mallampati, Intubation grade, BMI and type of medication.

A specific data collection form will be developed and the data will be collected retrospectively from patient journals.

The number is calculated to: n = 588, n = 294 before and after the implementation of PAC. We use a significance level of 5%. To achieve statistical strength of 80% (beta = 20%), we need 288 patients before and after PAC to detect a difference of at least 10%. Given that we have the opportunity to include many more then we assume that our study has adequate strength. Prevalences of cancellations are estimated as shares and presented with 95% confidence intervals (CIs) calculated using the exact method. Possible differences in background variables in patients included before and after the implementation of PAC will be estimated using kji-square tests or t-tests. The effect of the implementation of PAC will be estimated using logistic regression adjusted for possible confounding factors and results will be presented as adjusted odds ratio (OR) with 95% CI.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old.
* Open or laparoscopic surgery on elective patients after partial excision of the intestine.
* Patients following the ERAS (Enhanced recovery after surgery) protocol after the year 2014.
* Patients who attended PAC after the year 2017 and were assessed by anesthesia staff.

Exclusion Criteria:

* Emergency patients

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who have been to surgery for open or laparoscopic partial excision of the intestine.
Sampling Method: Non-Probability Sample
Enrollment: 2600 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-02-03 (Estimated); Study Completion 2027-04-03 (Estimated)

PRIMARY OUTCOMES:
Cancellation rate, Intraoperative events | 2014-2022
  Incidence of Cancellation rate and unanticipated intraoperative events

SECONDARY OUTCOMES:
Patient's characteristics , cancellation main events and concequenses. | 2014-2022
  Patients'characteristics, main events leading to cancellations of surgery, consequenses the cancellations brings to patients and the hospital.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kristoffersen EW, Fossum M, Tveit TO, Berge GT, Hagen MC, Opsal A. Comparison of elective hemicolectomy patients before and after establishment of a preoperative anaesthesia assessment clinic: a retrospective, observational study in a hospital in Norway. BMJ Open. 2025 Jun 12;15(6):e100922. doi: 10.1136/bmjopen-2025-100922. PMID 40506071